CLINICAL TRIAL: NCT05591677
Title: D-Cycloserine Augmentation of Intermittent Theta Burst Stimulation (iTBS) in Depression: A Multi-Site, Randomised, Placebo-Controlled Trial (COGENT)
Brief Title: D-Cycloserine Augmentation of Intermittent Theta Burst Stimulation (iTBS) in Depression (COGENT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Blue Bell Health, Australia (Unknown); Gold Coast Hospital and Health Service (Other Government)
Responsible Party: Principal Investigator, Leo Chen, Head, Clinical TMS and Psychopharmacology Research Units, Monash Alfred Psychiatry Research Centre (MAPrc), The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 567-22
Record Dates: First submitted 2022-10-16; First posted 2022-10-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active iTBS + active DCS 50mg/day (Active Comparator): Active iTBS (600 pulses), 5 days/week x 4 weeks + active DCS 50mg/day x 2 weeks, taken 2-hours prior to scheduled iTBS treatment.
  Interventions: Drug: D-Cycloserine; Device: Intermittent Theta Burst Stimulation
- Active iTBS + active DCS 100mg/day (Active Comparator): Active iTBS (600 pulses), 5 days/week x 4 weeks + active DCS 100mg/day x 2 weeks, taken 2-hours prior to scheduled iTBS treatment.
  Interventions: Drug: D-Cycloserine; Device: Intermittent Theta Burst Stimulation
- Active iTBS + placebo (Placebo Comparator): Active iTBS (600 pulses), 5 days/week x 4 weeks + placebo x 2 weeks, taken 2-hours prior to scheduled iTBS treatment.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Drug: D-Cycloserine — D-cycloserine (DCS) is a partial NMDA receptor agonist that has demonstrable impact on rTMS and TBS's neuromodulatory effects. Participants will be asked to orally ingest one capsule 2-hours prior to their scheduled iTBS treatment time.
  Arms: Active iTBS + active DCS 100mg/day; Active iTBS + active DCS 50mg/day
Device: Intermittent Theta Burst Stimulation — Intermittent Theta Burst Stimulation (iTBS) will be administered with a magnetic stimulator using a figure-of-8 coil or equivalent FDA-approved device. Initial treatment coil localisation and individual calibration of stimulation intensity will be conducted by TMS-trained investigators/staff using standard approaches.67,68 Stimulation intensity will be at 90% of the individual's calibrated resting motor threshold. iTBS treatment session delivers 600 pulses and is approximately 3½ minutes in duration. The total pulse number applied over a course of 20 treatments will be 12,000. This regimen is analogous with the iTBS protocol approved by the US FDA to treat TRD.

SUMMARY:
The goal of this clinical trial is to investigate if the drug D-Cycloserine (DCS) improves the antidepressant effects of Intermittent Theta Burst Stimulation (iTBS), a non-invasive brain stimulation therapy, in patients with Major Depressive Disorder (MDD). The main questions it aims to answer are:

* Whether taking DCS prior to iTBS therapy will be more effective in improving depressive symptoms than iTBS therapy alone.
* Compare the effect of DCS 100mg/day versus 50mg/day on depressive symptoms.
* Test the safety and tolerability of DCS. Participants will take either 50mg DCS per day, 100mg DCS or placebo prior to each iTBS treatment session. iTBS treatment will be administered daily, 5 days a week for 4 weeks. Clinical measures will be conducted at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a common and debilitating condition with high rates of treatment resistance. Repetitive transcranial magnetic stimulation (rTMS) is an established treatment for treatment-resistant depression with few adverse effects. Intermittent Theta Burst Stimulation (iTBS) is a time-efficient form of rTMS with evidence base in the treatment of treatment-resistant depression (TRD). The most commonly supported understanding of iTBS's mechanism of action appear to be its strengthening of connections between networks of neurons, which is modulated by the N-methyl-D-aspartate (NMDA) receptor. D-cycloserine (DCS) is a partial NMDA receptor agonist that has demonstrable impact on rTMS and TBS's neuromodulatory effects. This study protocol proposes the conduct of a prospective multi-site, parallel-arm design, randomized, double-blinded, placebo-controlled clinical trial to investigate DCS augmentation of iTBS in MDD. We will investigate if adjuvant DCS 50mg or 100mg/day might have superior iTBS antidepressant augmentation effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive episode (MDE), in accordance with the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5), in the context of unipolar major depressive disorder or bipolar affective disorder.
* 18 years or older in age.
* Treatment resistant depression at Stage II of the Thase and Rush classification.56
* Baseline Montgomery Åsberg Depression Rating Scale score of ≥ 20 (moderate-to-severe depression severity).57,58
* No increase or initiation of new antidepressant therapy in the four weeks prior to screening.
* Demonstrated capacity to give informed consent.

Exclusion Criteria:

* Inability to provide informed consent.
* Medically unstable patients at the discretion of the investigator.
* Concomitant neurological disorder or a history of a seizure disorder.
* Participants who are pregnant.
* Current substance use meeting DSM-5 criteria for substance use disorder.
* Per DSM-5, had ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder or delusional disorder as assessed by the Mini-International Neuropsychiatric Interview (MINI) at the time of screening.
* Diagnosis of any other mental disorder that is the participant's primary diagnosis or main mental health syndrome of concern at the time of screening, which may significantly affect psychiatric status and assessed as likely to impact trial participation, in the clinical judgement of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment response as per Montgomery Åsberg Depression Rating Scale (MADRS) | Determined at Week 4 (primary study endpoint)
  Clinical treatment response defined as >/= 50% reduction in MADRS scores from baseline to primary study endpoint.
  Clinician-administered depression rating scale. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.

SECONDARY OUTCOMES:
Change in Montgomery Åsberg Depression Rating Scale (MADRS) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Clinician-administered depression rating scale. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Change in Clinical Global Impression (CGI) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Clinician assessment of overall illness severity and global functioning. The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'. The CGI-Improvement scale is also rated 1-7, representing the range between 'Very much improved' and 'Very much worse'.
Change in Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Self-reported symptom rating scale for depression severity. Severity of depression can be judged based on the total score. 1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression.
Beck's Anxiety Inventory (BAI) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Self-reported symptom rating scale for anxiety severity. The score range is 0-63. A total score of 0-7 is considered minimal range, 8-15 is mild, 16-25 is moderate, and 26-63 is severe.
International Trauma Questionnaire (ITQ) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Self-reported symptom rating of trauma-related symptoms and their severity. All ITQ items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely).
Beck's Scale for Suicide Ideation (BSS) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Self-reported symptom rating scale for suicidal ideation. Scores range from 0 to 38, a higher score indicating a higher level of suicide ideation.
Change in World Health Organization Quality of Life (WHOQOL-BREF) | Administered at baseline and at the ends of weeks 1, 2, 3 and 4 of treatment.
  Self-reported rating scale of quality of life. Domains scores are calculated to range from 0-20 and scaled in a positive direction (ie. higher scores denote higher quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Leo Chen, MBBS PhD FRANZCP, Principal Investigator — The Alfred
Locations (1):
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No